CLINICAL TRIAL: NCT04794439
Title: Plaque Removal Efficacy of Four Dentifrices Following a Single Brushing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ST-20-U81
Record Dates: First submitted 2021-02-14; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque | interventions — Dentifrices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Toothpaste 1 with Stannous Fluoride (Active Comparator): Toothpaste with Stannous Fluoride
  Interventions: Drug: Dentifrices
- Toothpaste 1 with Sodium Fluoride and sodium bicarbonate (Active Comparator): Toothpaste with Sodium Fluoride and sodium bicarbonate
  Interventions: Drug: Dentifrices
- Toothpaste 2 with Stannous Fluoride (Active Comparator): Toothpaste with Stannous Fluoride
  Interventions: Drug: Dentifrices
- Toothpaste 2 with sodium Fluoride and sodium bicarbonate (Active Comparator): Toothpaste with sodium Fluoride and sodium bicarbonate
  Interventions: Drug: Dentifrices

INTERVENTIONS:
Drug: Dentifrices — Dentifrice on plaque

SUMMARY:
The purpose of this study is to evaluate and compare plaque removal efficacy of four dentifrices following a single timed tooth brushing. Prior to each evaluation visit of the four-way cross-over study, subjects will abstain from all oral hygiene for 24 hours. At each evaluation visit, subjects will be given a pre-brushing plaque evaluation, followed by a 1-minute supervised brushing and a post-brushing plaque evaluation.

DETAILED DESCRIPTION:
This study is a randomized, single-brushing, examiner-blinded, 4-cell cross-over design that enrolled approximately 70 subjects to ensure that at least 60 subjects to complete the study. This 4-week cross-over study will evaluate plaque removal following a single brushing with the assigned dentifrices. Qualified subjects will have sufficient plaque (Lobene-Soparkar Modification of Turesky Plaque Index). Subjects will be given a pre-brushing plaque evaluation, followed by a 1-minute supervised brushing and a post-brushing plaque evaluation.

ELIGIBILITY:
Inclusion Criteria:

1) 18 to 69 years

Exclusion Criteria:

1. Have any known allergies or sensitivities to marketed dentifrice or oral hygiene products.
2. Have fixed or removable orthodontic appliances, peri/oral piercings, or removable partial dentures.
3. Evidence of poor oral hygiene, rampant dental caries, presence of extrinsic stain or calculus deposits that may interfere with plaque assessments.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline (pre-brushing to post-brushing) in plaque score after single supervised use based on all surfaces of the whole mouth measured. | up to 4 weeks
  plaque evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No